CLINICAL TRIAL: NCT06767488
Title: Breathomics in the Diagnosis and Prediction of Radiotherapy-Induced Oropharyngeal Mucositis in Head and Neck Tumors
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-581
Record Dates: First submitted 2024-12-15; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Tumors; Breathomics; Volatile Organic Compounds; Radiotherapy-induced Oral Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — exhaled breath samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy-Induced Oropharyngeal Mucositis (RIOM) is one of the most distressing side effects for patients with head and neck tumors during radiotherapy, requiring clinical physicians to manage it according to the severity of mucositis to alleviate symptoms and improve quality of life. However, traditional diagnosis of RIOM overly relies on subjective evaluation, lacks early sensitivity, and existing biomarker diagnostic methods suffer from insufficient efficacy, invasiveness, and inconsistent results. This study aims to explore the diagnostic and predictive value of exhaled breathomics in RIOM of head and neck tumors. By collecting exhaled breath samples from head and neck tumor patients undergoing radiotherapy and analyzing volatile organic compounds (VOCs) using breath detection technology, we aim to develop and validate a non-invasive diagnostic and predictive model based on exhaled breathomics. The study will identify specific VOCs as potential biomarkers, providing new tools for early diagnosis, timely prediction, and personalized treatment of RIOM.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent. Over 18 years of age. Histologically confirmed head and neck tumors, treated with radiotherapy or chemoradiotherapy.

ECOG PS Score: 0/1/2.

Exclusion Criteria:

* Lung disease such as lung cancer, tuberculosis, and lung infections. Inhalation anesthesia within 3 months. Inhalation medication within 3 months. Postoperative laryngeal cancer. Concurrent serious uncontrolled medical conditions such as unstable heart disease requiring treatment, poorly controlled diabetes mellitus (fasting blood glucose > 1.5 x upper limit of normal).

Participation deemed inappropriate in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck tumors requiring radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Different grades radiotherapy-induced oral mucositis | Through study completion, up to 1 year
  The incidence rates of radiation-induced oral mucositis across various severity grades will be determined.

SECONDARY OUTCOMES:
Start and duration of radiotherapy-induced oral mucositis | Through study completion, up to 1 year
  Calculated the onset time and duration of radiotherapy-induced oral mucositis.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Southern medical university, Guangzhou, Guangdong, China